CLINICAL TRIAL: NCT03811184
Title: Validation of a Smartphone Application for the Assessment of Patients With Mild Cognitive Impairment: MemScreen
Acronym: MemScreen
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: MemScreen (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-A02672-53
Record Dates: First submitted 2019-01-17; First posted 2019-01-22 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-01

CONDITIONS: Cognitive Impairment; Alzheimer Disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MemScreen: Each participants will undergo MemScreen : a screening tool on smartphone for detecting mild cognitive impairment.
  Interventions: Diagnostic Test: MemScreen

INTERVENTIONS:
Diagnostic Test: MemScreen — Neuropsychological test on smartphone or digital tablet, on self assesment.

SUMMARY:
The clinical evaluation of a patient with a cognitive complaint requires neuropsychological tests, evaluating the integrity of memory and other cognitive functions.

The initial evaluation is made most often by a doctor (general practitioner). In case of need for further examination, a neuropsychological report is made in consultation memory by a neuropsychologist, with further cognitive tests.

The Cognitive Neurology Center at Lariboisière Hospital - Fernand Widal has developed a tool on a digital tablet or smartphone to evaluate cognitive functions: MemScreen.

The purpose of this study is to validate this new neuropsychological test on tablet compared to the neuropsychological reference tests.

DETAILED DESCRIPTION:
Characteristics of MemScreen :

* Smartphone / tablet application developed by the Cognitive Neurology Center at Lariboisière - Fernand Widal Hospital to explore a patient with a cognitive disorder.
* The application is a self-test by the patient under the supervision of a doctor.
* The doctor has an account to be able to pass the test to patients.
* The tablet test is anonymous without the possibility to identify the patient.

ELIGIBILITY:
Inclusion Criteria:

* Major patients followed in memory clinic.
* Performing a neuropsychological assessment less than 6 months old.
* No visual or motor deficiency impeding the use of a digital tablet.

Exclusion Criteria:

* None.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population seen on memory clinic for memory complaints.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-01-17 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Ability to detect patients with mild cognitive impairment. | through study completion, an average of 6 months
  To evaluate the ability of MemScreen to discriminate patients with an objective memory disorder from a validated neuropsychological reference test: the free and cued selective reminding test.

CONTACTS AND LOCATIONS:
Overall Officials: Julien Dumurgier, MD, Principal Investigator — Cognitive Neurology Center of Lariboisiere Hospital
Locations (1):
- Centre Neurologie Cognitive Hôpital Fernand Widal, Paris, France

IPD SHARING:
Plan to Share IPD: No